CLINICAL TRIAL: NCT04874467
Title: Influence of Keratinized Mucosa on Dental Implants With Mucositis in Patients Undergoing Supportive Periodontal Therapy
Brief Title: Influence of Keratinized Mucosa on Dental Implants With Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Clinical Instructor, Universitat Internacional de Catalunya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PER-ECL-2020-02
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Compliance, Patient
MeSH Terms: conditions — Peri-Implantitis; Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keratinized Mucosa ≥ 2 mm (Experimental): Supportive periodontal therapy, in teeth by means of ultrasonic devices and manual curettes. In implants using the same devices but made of titanium. Oral hygiene instructions
  Interventions: Procedure: Supportive periodontal therapy
- Keratinized Mucosa < 2 mm (Experimental): Supportive periodontal therapy, in teeth by means of ultrasonic devices and manual curettes. In implants using the same devices but made of titanium. Oral hygiene instructions
  Interventions: Procedure: Supportive periodontal therapy

INTERVENTIONS:
Procedure: Supportive periodontal therapy — A complete professional prophylaxis session will be performed, which includes ultrasound debridement, scaling with curettes and dental polishing with a rubber cup. On the other hand, in implants affected by mucositis, supra and sub-gingival debridement will be performed using a combination of ultrasound with a titanium tip and titanium curettes.
  All patients will receive personalized hygiene instructions. Patients will be instructed to brush their implants twice daily using the modified Bass technique with a medium-hard manual toothbrush and low-abrasive toothpaste. In addition, they will be taught to use specific interproximal brushes. If access with an interdental brush is not possible, flossing will be indicated. Oral hygiene instructions will be reviewed at each visit.

SUMMARY:
Introduction:

It seems that some local and systemic factors can be associated with an increased incidence of peri-implant diseases. Predisposing to an increase inflammatory response when plaque is present.

There is still controversy on which factors can be considered as risk indicators. One of them is the keratinized mucosa width (KM), that seems to facilitate plaque control around implants.

Objectives:

Assess the relationship between keratinized mucosa and the recurrence of mucositis, comparing bleeding on probing (BOP) in implants with mucositis for 24 weeks after implant disinfection therapy, the control group is defined by having KM ≥ 2 mm and the test group KM < 2 mm.

Material and methods:

38 patients presenting one single implant each with a single screw retained crown loaded for at least 1 year. Periodontal maintenance therapy will be performed and oral hygiene instruction will be delivered. Follow up visits will be after 8, 12 and 24 weeks in which the following parameters will be registered: Keratinized Mucosa width, Attached mucosa, Gingival Index, Vestibule Depth, Mucosa Thickness. Probing Pocket Depth, Recession, modified Plaque Index, Bleeding on Probing, modified Bleeding Index. Also a microbiologic test will be taken in the implant sulcus before the periodontal maintenance therapy and at 24 weeks.

A multilevel statistical analysis will be conducted comparing the control and the test group, adjusting for the correlation among multiple observations.

DETAILED DESCRIPTION:
Introduction:

It seems that some local and systemic factors can be associated with an increased incidence of peri-implant diseases. Predisposing to an increase inflammatory response when plaque is present.

There is still controversy on which factors can be considered as risk indicators. One of them is the keratinized mucosa width (KM), that seems to facilitate plaque control around implants.

Objectives:

Assess the relationship between keratinized mucosa and the recurrence of mucositis, comparing bleeding on probing (BOP) in implants with mucositis for 24 weeks after implant disinfection therapy, the control group is defined by having KM ≥ 2 mm and the test group KM < 2 mm.

Methods:

38 patients presenting one single implant each with a screw retained crown loaded for at least 1 year. Periodontal maintenance therapy will be performed and oral hygiene instruction will be delivered. Follow up visits will be after 8, 12 and 24 weeks in which the following parameters will be registered: Keratinized Mucosa width, Attached mucosa, Gingival Index, Vestibule Depth, Mucosa Thickness. Probing Pocket Depth, Recession, modified Plaque Index, Bleeding on Probing, modified Bleeding Index. Also a microbiologic test will be taken in the implant sulcus before the periodontal maintenance therapy and at 24 weeks.

A multilevel statistical analysis will be conducted comparing the control and the test group, adjusting for the correlation among multiple observations.

ELIGIBILITY:
Inclusion Criteria:

* patients> 18 years;
* smokers <10 cigarettes / day;
* partially edentulous patients. The spaces must be associated with at least one adjacent mesial and one distal tooth;
* presence of bleeding and / or suppuration on probing, erythema and inflammation;
* absence of radiographic bone loss around implant distance (<2mm from expected radiographic marginal bone level);
* individual dental implants rehabilitated for more than a year;
* screw-retained restorations on implants;
* absence of active periodontal disease;
* who have not taken systemic antibiotics in the last 3 months;
* adequate oral hygiene motivation and collaboration defined as plaque index <25%

Exclusion Criteria:

* totally edentulous patients;
* uncontrolled systemic diseases;
* diseases of the mucosa (erosive lichen planus, etc.);
* taking medications that may interfere with periodontal health or healing; (corticosteroids, calcium channel antagonists, antiepileptic drugs, immunosuppressants, etc.)
* pregnant or lactating patients;
* cemented implant restorations;
* restorations on implants over contoured that cannot be corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 24 weeks
  The main objective of the study is to evaluate the association between MQ and recurrence of mucositis, comparing the bleeding index on probing (BoP) in implants that have mucositis, in a control group characterized by 2 mm or more of MQ and a test group characterized by less than 2 mm of MQ over a 24-week period after peri-implant maintenance therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, DDS PhD, Study Chair — Universitat Internacional de Catalunya
Locations (1):
- International University of Catalunya, Barcelona, Spain

REFERENCES:
- [Derived] Blasi G, Chierico F, Amerio E, Alvarez G, Isabal S, Arredondo A, Blanc V, Nart J, Monje A. Influence of keratinized mucosa width on the resolution of peri-implant mucositis: A prospective cohort study. Clin Implant Dent Relat Res. 2024 Jun;26(3):581-591. doi: 10.1111/cid.13317. Epub 2024 Mar 1. PMID 38426741